CLINICAL TRIAL: NCT05656170
Title: Pre-Operative Stellate Ganglion to Prevent Post-Operative Atrial Fibrillation
Brief Title: Stellate Ganglion to Prevent Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to begin study
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21022602
Record Dates: First submitted 2021-05-07; First posted 2022-12-19 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation New Onset
Keywords: post-operative arrhythmias; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stellate ganglion block arm (Experimental): This arm will receive a one time bilateral stellate ganglion block with 20 cc bupivacaine (10 cc per side).
  Interventions: Procedure: Stellate ganglion block; Drug: Bupivacain
- Placebo arm (Sham Comparator): This arm will receive a one time bilateral injection with 20 cc normal saline(10 cc per side).
  Interventions: Procedure: Stellate ganglion block; Drug: Saline

INTERVENTIONS:
Procedure: Stellate ganglion block — Ultrasound will be utilized to identify anatomic landmarks and prepare for the stellate ganglion block. Skin will be prepped with chloraprep. The C6 level is identified. The Chassaignac tubercle (the anterior tubercle of the C6 vertebral body) is then identified. Placement of the ultrasound transducer helps retract the carotid sheath and sternocleidomastoid muscle laterally. Pressure is applied with the ultrasound transducer to reduce the distance between the skin and tubercle.
  The needle is inserted towards to the Chassaignac tubercle after contact it is redirected towards the body of C6. The needle is then withdrawn 1-2 mm to bring it out of the longus colli muscle while still staying within the prevertebral fascia. After negative aspiration, 1-2 mL of local anesthetic (or normal saline in the placebo group) is injected, and spread can be visualized with ultrasound. Once confirming that the injection was subfascial, the remaining local anesthetic can be given (10 mL in total).
Drug: Bupivacain — The intervention group will receive bupivacaine injection guided by ultrasound at the location of the stellate ganglion.
  Arms: Stellate ganglion block arm
Drug: Saline — The control group will receive a normal saline injection guided by ultrasound at the location of the stellate ganglion.
  Arms: Placebo arm

SUMMARY:
New onset atrial fibrillation is a common problem after cardiac surgery. The reported incidence after coronary artery bypass grafting (CABG) is 15-40%, 37-50% after valve surgery, and up to 60% after CABG and valve surgery. Post-operative atrial fibrillation (POAF) is associated with increase risk for stroke, increased length of hospital stay, increase risk of other new arrhythmias, increased need for pacemaker implantation, and increased mortality. Several interventions have been implemented in order to prevent post-operative atrial fibrillation including use of betablockers, sotalol, amiodarone, atrial pacing, and antioxidant vitamins. Despite these interventions (several carry risk of adverse effects) POAF remains common.

Cardiac sympathetic innervation arises from the stellate ganglion. Stellate ganglion block (SGB) with local anesthetic agents (lidocaine or bupivacaine) can reduce sympathetic output to the heart with minimal side effects. This procedure has been successfully utilized in patients with medication refractory ventricular arrhythmias. In atrial tissue SGB has been shown to prolong atrial effective refractory periods, reduce atrial arrhythmia inducibility, and shorten atrial fibrillation duration in patients who have atrial fibrillation. Pre-operative SGB has been utilized to prevent post-operative radial artery spasm (when the radial artery was used a coronary bypass graft conduit). The investigators hypothesize that pre-operative SGB will reduce the incidence of post-operative new atrial fibrillation in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Post-operative atrial fibrillation (POAF) is a widely recognized problem after cardiac surgery. Atrial fibrillation is the most common arrhythmia to occur after cardiac surgery. The reported incidence after coronary artery bypass grafting (CABG) is 15-40%, 37-50% after valve surgery, and up to 60% after CABG and valve surgery1-3. Most POAF episodes occur by day three2. Postoperative AF is associated with increased risk of postoperative stroke (3.3% versus 1.4%), increased length of hospital stay (ICU stay 5.7 versus 3.4 days, floor stay 10.9 versus 7.5 days), increased incidence of ventricular arrhythmias (9.2% versus 4.0%), increased need for permanent pacemaker implant (3.7% versus 1.6%), and increased mortality3-5.

Multiple therapies have been proposed to prevent POAF in order to reduce hospital length of stay and possibly the risk of stroke and death. Beta blockers, sotalol, amiodarone, atrial pacing, and antioxidant vitamins have all been shown to lower risk of POAF6-11. Beta blockers are the most frequently used medications owning to safety, ease of use, cost-effectiveness, and familiarity. Long-term beta blocker therapy is indicated in many patients undergoing cardiac surgery anyway due to underlying cardiac conditions (coronary artery disease, cardiomyopathy, etc). The other interventions are associated with increased adverse effects and/or unclear added benefit in addition to beta blockers12.

Cardiac sympathetic innervation arises from the stellate ganglion. The stellate ganglia can be temporarily anesthetized by percutaneous injection of local anesthetic (such as lidocaine, bupivacaine, or ropivacaine). This procedure can be done at bedside with ultrasound guidance. Stellate ganglion block (SGB) can reduce sympathetic output to the heart with minimal system effect. The post ganglionic fibers from the stellate ganglion release not only norepinephrine (the target of beta blockers) but several additional neurotransmitters (including neuropeptide Y and galanin) that modulate adrenergic signaling13,14. SGB provides added benefit in addition to both beta blockers and antiarrhythmics (such as amiodarone) for the suppression of refractory ventricular tachycardia15. The effect of SGB on arrhythmia suppression can last up to several weeks, the longer duration of efficacy relative to drug half-life is likely due to alterations in neuro-transmission and neural processing.

While SGB has been most widely applied to refractory ventricular arrhythmias, there are antiarrhythmic effects in the atrial also. In a canine model stellate ganglion stimulation facilities AF induction and worsened atrial electrical properties (shortened atrial effective refractory period (ERP) and increased dispersion of the atrial ERP). SGB reduced AF initiation16. This effect is similar in humans; SGB prolongs atrial ERP, reduces atrial inducibility, and in those with inducible AF, shortens AF duration17. One study evaluating pre-operative SGB to reduce the risk of radial artery spasm when the radial artery was used as a coronary bypass conduit found a significantly lower incidence of post-operative atrial fibrillation, inotropic agent use, and ST segment depression in those who received SGB18. SGB may have a similar or complimentary effect to low level vagal nerve stimulation, which has been shown to reduce POAF in cardiac surgery patients19.

B. OBJECTIVES

Hypothesis:

Pre-operative stellate ganglion block, in addition to beta blockade, will reduce post-operative atrial fibrillation in cardiac surgery patients.

Specific aims:

Primary end point: Incidence of new onset atrial fibrillation after CABG surgery Secondary end points: atrial fibrillation burden (time spent in atrial fibrillation), incidence of any arrhythmia, occurrence of any adverse effects from the stellate block.

STUDY DESIGN

a. Study design: Single-blind placebo-controlled study. Patients will be randomized at the time of their preoperative surgical visit to either stellate ganglion block with 1% lidocaine or 0.25% bupivacaine versus saline injection. Patients will remain blinded to their treatment allocation. Both treatment options will use standard-of-care surgical approach and techniques. The distinction is only in the allocation toward stellate ganglion block versus saline injection. Cross-over is not anticipated to occur.

Surgical procedure will be per routine surgical practice in accordance with the standard of care.

After surgery all patients will be monitored with standard cardiac telemetry monitors in accordance with current standard of care. Cardiac rhythm will be reviewed up to the day of discharge in order to identify the occurrence of atrial fibrillation and document burden of atrial fibrillation. If atrial fibrillation occurs, it will be treated in accordance with current standard of care practices.

Duration of study: 24 months Randomization scheme: patients will be allocated in a 1 to 1 fashion using to stellate ganglion block versus saline injection at the time of their pre-surgical appointment.

STUDY PROEDURES

Pre-procedure:

* Patients will be screened for the study
* A written informed consent will be obtained
* Patients will be randomized in a 1 to 1 fashion to either stellate ganglion block with 1% lidocaine or saline injection Stellate ganglion block After the patient is placed under general anesthesia ultrasound will be utilized to identify anatomic landmarks and prepare for the stellate ganglion block. Skin will be prepped with chloraprep. The needle insertion site is located between the trachea and the carotid sheath. The C6 level is identified at the level of the cricoid cartilage. The Chassaignac tubercle (the anterior tubercle of the C6 vertebral body) is then identified. Placement of the ultrasound transducer helps retract the carotid sheath and sternocleidomastoid muscle laterally. Pressure is applied with the ultrasound transducer to reduce the distance between the skin and tubercle.

The needle is inserted towards to the Chassaignac tubercle, and, after contact, it is redirected inferomedially towards the body of C6. The needle is then withdrawn 1-2 mm to bring it out of the longus colli muscle while still staying within the prevertebral fascia. After negative aspiration, 1-2 mL of local anesthetic can be injected, and spread can be visualized with ultrasound. Once confirming that the injection was subfascial, the remaining local anesthetic can be given (10 mL in total).

The patient will be assessed for Horner syndrome (ptosis, miosis, anhidrosis) and skin temperature will be monitored to identify a skin temperature increase greater than 3°F. A dry dressing can be placed over puncture site if needed.

After surgery patients will be monitored in the cardiac surgery intensive care unit per usual practice. All patients will be monitored with standard hospital continuous cardiac telemetry. Telemetry data will be reviewed to identify new onset atrial fibrillation and to document atrial fibrillation burden.

STATISTICAL PLAN AND CONSIDERATIONS

Sample size estimation:

The sample size for this study is a total of 80 subjects (40 stellate ganglion block and 40 control). The sample size estimate was based on a goal to observe an absolute 50% difference in the incidence of post-operative atrial fibrillation between the two groups, leading to a Cohen's d statistic of 1. With a significance level (α) = 0.05 and a power of 0.8, at least 31 subjects will be required in each group.

Statistical methods:

Patients will be studied based on the final treatment allocation. Fisher's exact or the Chi-Square test will be used for categorical variables, and continuous parameters will be compared by the two-tailed unpaired Student's t test and the F test for analysis of variance (ANOVA), as needed.

RISKS AND BENEFITS There are risks with stellate ganglion block which include, but are not limited to, the risk of infection, injury to adjacent vascular structures (resulting in hematoma formation), inadvertent intravascular or intrathecal injection, anesthesia of the recurrent laryngeal nerve (can produce temporary hoarseness), anesthesia of the phrenic nerve (can result in temporary elevated hemidiaphragm), pneumothorax, esophageal perforation, chylothorax, bradycardia, hypotension, and heart block. The use of real time ultrasound guidance can minimize risk.

Benefits include possible reduction in the risk of post-operative atrial fibrillation and other cardiac arrhythmias.

SAFETY AND ADVERSE EVENTS

Safety:

Periprocedural complications will be logged. Complications will be independently reviewed at the midpoint by the site's primary investigator. Should there be a trend towards increased complication risk, the study will be halted.

Adverse Events:

As noted above, all adverse events associated with the stellate ganglion block will be monitored periprocedurally and continuously through the study.

DATA HANDLING AND RECORD KEEPING Data will be collected on paper by study coordinators and transcribed into an electronic database which will be maintained on-campus locations at RUMC. Data will be managed by the PIs and study coordinators. Access to the data will be limited to study investigators and research coordinators only during the study enrollment period.

All patient specific identifiers will be kept separate from the primary research database. The research database will be organized by a unique patient identifier.

STUDY MONITORING, AUDITING AND INSPECTING All periprocedural complications and adverse events will be reviewed by the investigators at study midpoint to ensure there is no significant difference in event rate between the study groups. Should there be significant differences, or if there should be a high overall event-rate out-of-line with the procedural norm, the study will be halted.

FINANCIAL CONSIDERATIONS No remuneration will be provided to subjects.

ETHICAL CONSIDERATIONS No specific ethical considerations are identified in relation to this study.

CONFLICT OF INTEREST None.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old scheduled to undergo elective coronary artery bypass (CABG) surgery based on current surgical guidelines.

Exclusion Criteria:

* Prior history of atrial fibrillation
* Current antiarrhythmic use (other than beta blockers)
* Inability of patient to provide consent for themselves either due to medical or psychiatric comorbidity
* Non-elective surgery
* Patients undergoing mitral valve replacement or repair surgery
* Patients undergoing surgical MAZE procedure
* Pregnancy
* History of neck surgery
* Systemic or local infection
* Current coagulopathy
* Pathologic bradycardia (baseline heart rate <50 beats/minute or untreated atrioventricular block)
* History of glaucoma
* Allergy to lidocaine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of new onset atrial fibrillation after CABG surgery | from surgery completion to discharge, up to 1 month
  Atrial fibrillation will be identified by Continuous cardiac rhythm monitoring (telemetry) throughout the post operative period

SECONDARY OUTCOMES:
Duration of atrial fibrillation | from surgery completion to discharge, up to 1 month
  Total time in atrial fibrillation will be recorded from Continuous cardiac rhythm monitoring (telemetry)
Incidence of any other arrhythmias (such as atrial flutter, atrial tachycardia, premature ventricular contractions, or ventricular tachycardia) | from surgery completion to discharge, up to 1 month
  Continuous cardiac rhythm monitoring (telemetry) will be reviewed throughout the post-operative admission

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Larsen, DO, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maisel WH, Rawn JD, Stevenson WG. Atrial fibrillation after cardiac surgery. Ann Intern Med. 2001 Dec 18;135(12):1061-73. doi: 10.7326/0003-4819-135-12-200112180-00010. PMID 11747385
- [Background] Mathew JP, Fontes ML, Tudor IC, Ramsay J, Duke P, Mazer CD, Barash PG, Hsu PH, Mangano DT; Investigators of the Ischemia Research and Education Foundation; Multicenter Study of Perioperative Ischemia Research Group. A multicenter risk index for atrial fibrillation after cardiac surgery. JAMA. 2004 Apr 14;291(14):1720-9. doi: 10.1001/jama.291.14.1720. PMID 15082699
- [Background] Creswell LL, Schuessler RB, Rosenbloom M, Cox JL. Hazards of postoperative atrial arrhythmias. Ann Thorac Surg. 1993 Sep;56(3):539-49. doi: 10.1016/0003-4975(93)90894-n. PMID 8379728
- [Background] Kosmidou I, Chen S, Kappetein AP, Serruys PW, Gersh BJ, Puskas JD, Kandzari DE, Taggart DP, Morice MC, Buszman PE, Bochenek A, Schampaert E, Page P, Sabik JF 3rd, McAndrew T, Redfors B, Ben-Yehuda O, Stone GW. New-Onset Atrial Fibrillation After PCI or CABG for Left Main Disease: The EXCEL Trial. J Am Coll Cardiol. 2018 Feb 20;71(7):739-748. doi: 10.1016/j.jacc.2017.12.012. PMID 29447735
- [Background] Mariscalco G, Klersy C, Zanobini M, Banach M, Ferrarese S, Borsani P, Cantore C, Biglioli P, Sala A. Atrial fibrillation after isolated coronary surgery affects late survival. Circulation. 2008 Oct 14;118(16):1612-8. doi: 10.1161/CIRCULATIONAHA.108.777789. Epub 2008 Sep 29. PMID 18824644
- [Background] Crystal E, Connolly SJ, Sleik K, Ginger TJ, Yusuf S. Interventions on prevention of postoperative atrial fibrillation in patients undergoing heart surgery: a meta-analysis. Circulation. 2002 Jul 2;106(1):75-80. doi: 10.1161/01.cir.0000021113.44111.3e. PMID 12093773
- [Background] Arsenault KA, Yusuf AM, Crystal E, Healey JS, Morillo CA, Nair GM, Whitlock RP. Interventions for preventing post-operative atrial fibrillation in patients undergoing heart surgery. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003611. doi: 10.1002/14651858.CD003611.pub3. PMID 23440790
- [Background] Burgess DC, Kilborn MJ, Keech AC. Interventions for prevention of post-operative atrial fibrillation and its complications after cardiac surgery: a meta-analysis. Eur Heart J. 2006 Dec;27(23):2846-57. doi: 10.1093/eurheartj/ehl272. Epub 2006 Oct 2. PMID 17015402
- [Background] Harling L, Rasoli S, Vecht JA, Ashrafian H, Kourliouros A, Athanasiou T. Do antioxidant vitamins have an anti-arrhythmic effect following cardiac surgery? A meta-analysis of randomised controlled trials. Heart. 2011 Oct;97(20):1636-42. doi: 10.1136/heartjnl-2011-300245. Epub 2011 Aug 23. PMID 21865202
- [Background] Mitchell LB, Exner DV, Wyse DG, Connolly CJ, Prystai GD, Bayes AJ, Kidd WT, Kieser T, Burgess JJ, Ferland A, MacAdams CL, Maitland A. Prophylactic Oral Amiodarone for the Prevention of Arrhythmias that Begin Early After Revascularization, Valve Replacement, or Repair: PAPABEAR: a randomized controlled trial. JAMA. 2005 Dec 28;294(24):3093-100. doi: 10.1001/jama.294.24.3093. PMID 16380589
- [Background] Herring N, Cranley J, Lokale MN, Li D, Shanks J, Alston EN, Girard BM, Carter E, Parsons RL, Habecker BA, Paterson DJ. The cardiac sympathetic co-transmitter galanin reduces acetylcholine release and vagal bradycardia: implications for neural control of cardiac excitability. J Mol Cell Cardiol. 2012 Mar;52(3):667-76. doi: 10.1016/j.yjmcc.2011.11.016. Epub 2011 Dec 7. PMID 22172449
- [Background] Herring N, Lokale MN, Danson EJ, Heaton DA, Paterson DJ. Neuropeptide Y reduces acetylcholine release and vagal bradycardia via a Y2 receptor-mediated, protein kinase C-dependent pathway. J Mol Cell Cardiol. 2008 Mar;44(3):477-85. doi: 10.1016/j.yjmcc.2007.10.001. Epub 2007 Oct 11. PMID 17996892
- [Background] Meng L, Tseng CH, Shivkumar K, Ajijola O. Efficacy of Stellate Ganglion Blockade in Managing Electrical Storm: A Systematic Review. JACC Clin Electrophysiol. 2017 Sep;3(9):942-949. doi: 10.1016/j.jacep.2017.06.006. PMID 29270467
- [Background] Zhou Q, Hu J, Guo Y, Zhang F, Yang X, Zhang L, Xu X, Wang L, Wang H, Hou Y. Effect of the stellate ganglion on atrial fibrillation and atrial electrophysiological properties and its left-right asymmetry in a canine model. Exp Clin Cardiol. 2013 Winter;18(1):38-42. PMID 24294036
- [Background] Leftheriotis D, Flevari P, Kossyvakis C, Katsaras D, Batistaki C, Arvaniti C, Giannopoulos G, Deftereos S, Kostopanagiotou G, Lekakis J. Acute effects of unilateral temporary stellate ganglion block on human atrial electrophysiological properties and atrial fibrillation inducibility. Heart Rhythm. 2016 Nov;13(11):2111-2117. doi: 10.1016/j.hrthm.2016.06.025. Epub 2016 Jun 21. PMID 27353237
- [Background] Yildirim V, Akay HT, Bingol H, Bolcal C, Iyem H, Doganci S, Demirkilic U, Tatar H. Pre-emptive stellate ganglion block increases the patency of radial artery grafts in coronary artery bypass surgery. Acta Anaesthesiol Scand. 2007 Apr;51(4):434-40. doi: 10.1111/j.1399-6576.2006.01260.x. PMID 17378781
- [Background] Stavrakis S, Humphrey MB, Scherlag B, Iftikhar O, Parwani P, Abbas M, Filiberti A, Fleming C, Hu Y, Garabelli P, McUnu A, Peyton M, Po SS. Low-Level Vagus Nerve Stimulation Suppresses Post-Operative Atrial Fibrillation and Inflammation: A Randomized Study. JACC Clin Electrophysiol. 2017 Sep;3(9):929-938. doi: 10.1016/j.jacep.2017.02.019. Epub 2017 May 30. PMID 29759717